CLINICAL TRIAL: NCT03910621
Title: A Single Arm Uncontrolled 12 Months Clinical Study to Evaluate the Safety and Efficacy of Miglustat (Zavesca) for the Treatment of Niemann Pick Type C Disease (NPC) in Chinese Subjects
Brief Title: Safety and Efficacy of Miglustat in Chinese NPC Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-056C405
Record Dates: First submitted 2019-03-08; First posted 2019-04-10 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Niemann-Pick Disease, Type C
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — miglustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Miglustat (Experimental): Miglustat is administered three times a day as an oral capsule
  Interventions: Drug: Miglustat

INTERVENTIONS:
Drug: Miglustat — capsule, oral use

SUMMARY:
This is a prospective, multi-center, open-label, non-randomized, single-arm Phase IV confirmatory study.

Approximately 19 subjects with Niemann Pick Type C disease (NPC) will be enrolled in this study. The study will be conducted at 2 sites in China.

DETAILED DESCRIPTION:
This is a prospective, multi-center, open-label, non-randomized, single-arm Phase IV confirmatory study.The study is conducted in Chinese subjects aged 4 years and older with Niemann Pick Type C disease (NPC). Approximately 19 subjects will be enrolled in this study. The study will be conducted at 2 sites in China. Patients will be treated with miglustat for 12 months, efficacy and safety outcomes will be measured

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed 2 pathogenic mutations in either Niemann Pick Type C Gene 1 or 2 (NPC 1 or NPC 2) or 1 pathogenic mutation in either NPC1 or NPC2 plus a positive biomarker (oxysterol or lysosphingolipids or bile acids) plus high clinical suspicion
* Signed informed consent prior to any study-mandated procedure.
* For subjects who are younger than 18 years consent must be sought of at least one legal guardian who shall sign the informed consent form and indicate the relationship between him/her and the subject.
* Subjects who are 18 years or older must sign the consent. If the subject cannot make an independent decision to participate in the study, consent must be sought of the legal agents who shall sign the informed consent form and indicate the relationship between him/her and the subject.
* Male and female subjects aged 4 years and older.
* Subjects who can performed the tests for the horizontal and vertical saccadic eye movements;
* Subjects who are able to swallow the study drug;
* Women of childbearing potential are only eligible if the following applies:
* Negative urine pregnancy test at screening.
* Agreement to undertake monthly urine pregnancy tests during the study and up to at least 30 days after study treatment discontinuation.
* Agreement to use one of the methods of birth control / follow the contraception scheme from screening up to at least 30 days after study treatment discontinuation.
* A fertile male (physiologically capable of fathering a child according to investigator's judgment) is eligible only if he agrees to use a condom during the treatment period and for an additional 12 weeks after treatment discontinuation.

Exclusion Criteria:

Subjects must not fulfill any of the following exclusion criteria. It is not permitted to waive any of the criteria for any subject:

* Subjects suffering from clinically significant diarrhea (>3 liquid stools per day for >7 days) without definable cause within 3 months before enrollment.
* Known hypersensitivity to the investigational treatment or drugs of the same class, or any of their excipients.
* Subjects who suffer from renal insufficiency with a creatinine clearance rate (CCR) of < 30ml/min per 1.73m2.
* Pregnant, planning to be become pregnant or lactating females, not using reliable birth control male adult subjects.
* Previous exposure to investigational treatment for more than 12 months before study start.
* Planned or current treatment with another investigational treatment up to 3 months prior to randomization. Symptomatic therapies are allowed (such as curcumin).
* Any known factor or disease that might interfere with treatment compliance, study conduct, or interpretation of the results, such as drug or alcohol dependence or psychiatric disease, end stage disease including wheelchair bound patients, bedridden patients etc.
* Subjects who are judged unqualified for the clinical trial by the investigator.
* Subjects who suffer lysosomal storage diseases, enzyme deficiency or neurological diseases other than NPC.
* Subjects who suffer variant filipin staining without confirmatory genetic diagnosis of NPC.
* Subjects with uncontrolled epilepsy.
* Subjects with complete ophthalmoplegia.
* Known concomitant life-threatening disease with a life expectancy < 12 months.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Observed change in HSEM (ms/deg) | baseline to week 52
  Change in HSEM from baseline to week 52

SECONDARY OUTCOMES:
Change in Pineda disability scale score | baseline to week 52
  Change in the modified Pineda disability scale score. The scale is assessing 4 key domains (manipulation, ambulation, language and swallowing). Individual scores of the domains are claculated ted into a composite score, 6 being the lowest and best score and 24 being the worst and highest score.
Incidence of treatment-emergent AEs and SAEs | Baseline to 30 days after End of Treatment (Week 52)
  Treatment-emergent adverse events (AEs) up to 30 days after EOT

CONTACTS AND LOCATIONS:
Overall Officials: Yue Wu, Study Director — Janssen China R&D
Locations (2):
- China (2):
  - Peking University first Hospital, Beijing
  - Xin Hua Hospital, Shanghai Jiao Tong University, Shanghai

REFERENCES:
- [Derived] Zhang H, Xiong H, Wei C, Yi M, Che Y, Zhuo J, Li X. Evaluation of the safety and efficacy of miglustat for the treatment of Chinese patients with Niemann-Pick disease type C: A prospective, open-label, single-arm, phase IV trial. Intractable Rare Dis Res. 2024 Nov 30;13(4):227-235. doi: 10.5582/irdr.2024.01056. PMID 39628618